CLINICAL TRIAL: NCT02706015
Title: National, Phase III, Multicenter, Randomized, Double-Blind, Parallel, Non-Inferiority Trial to Evaluate the Efficacy and Safety of Cefaliv® Compared to the Neosaldina® in the Treatment of Migraine Attacks
Brief Title: Cefaliv® Compared to Neosaldina® in the Treatment of Migraine Attacks
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic reasons of the company
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACH-CFL-03(10/14)
Record Dates: First submitted 2015-11-23; First posted 2016-03-11 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Migraine Headache
Keywords: Headache; Aura; Migraine
MeSH Terms: conditions — Migraine Disorders; Headache; Epilepsy | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cefaliv® & Placebo (Experimental): Dihydroergotamine mesylate+ dipyrone sodium + caffeine
  Interventions: Drug: Cefaliv® & Placebo
- Neosaldina® & Placebo (Active Comparator): Isometheptene mucate + dipyrone sodium + anhydrous caffeine
  Interventions: Drug: Neosaldina® & Placebo

INTERVENTIONS:
Drug: Cefaliv® & Placebo — 02 tablet of Cefaliv® + 02 tablet of comparator placebo, VO, after the beging of migraine with with mild to moderate pain
  Other Names: Cefaliv® (Dihydroergotamine mesylate+ dipyrone sodium + caffeine) & Placebo
  Arms: Cefaliv® & Placebo
Drug: Neosaldina® & Placebo — 02 tablets of Neosaldina® + 02 tablet of comparator placebo, VO, after the beging of migraine with with mild to moderate pain
  Other Names: Neosaldina® (Isometheptene mucate + dipyrone sodium + anhydrous caffeine) & Placebo
  Arms: Neosaldina® & Placebo

SUMMARY:
This study evaluates the non-inferiority of Cefaliv® compared to Neosaldina® in the treatment of migraine attack in two hundred and sixteen adults of both sexes with age between eighteen and sixty five years old. The first Half of participants will receive Cefaliv®, the other half will receive Neosaldina®.

DETAILED DESCRIPTION:
Cefaliv® is a combination of 3 drugs: dihydroergotamine mesylate, dipyrone sodium, and caffeine. The dihydroergotamine mesylate interacts with the serotonergic, dopaminergic and noradrenergic receptors, but it's mechanism is not totally known. The dipyrone is a non-steroidal antiinflammatory which has an analgesic, antiinflammatory and antipyretic effect. And the caffeine presents mechanisms that are not totally clear, but it may relieves the pain by activating of the central noradenosine pathway (pain suppressing system).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of both sexes;
2. Age older or equal to 18 and younger than 66 years if they have symptoms of migraine headache before 50 years of age;
3. Presence of migraine headache with or without aura symptoms, at least 03 months prior to the study, the criteria defined by International Classification of Headache Disorders(ICHD)-II, 2004 International Headache Society(IHS) - Annex I;
4. Subjects which are experiencing 2-6 migraine attacks per month with mild to moderate pain intensity in the last 3 months prior to screening visit;
5. Subjects which are able to distinguish migraine attacks to any other type of headache;
6. Aptitude to understand and consent to participate in this clinical study, manifested by signing the Informed Consent and Informed (IFC);

Exclusion Criteria:

1. Any clinical finding (clinical evaluation / physical) that is interpreted by the Investigator as a risk to the participant in the clinical trial;
2. Subjects which had recent episodes of headache, with frequency equal or higher than 15 daily episodes per month, 3 months prior to the screening visit;
3. Subjects with headache history defined by the ICHD-II criteria, 2004 IHS (International Headache Society) rated as:

   * Typical aura with non-migraine headache;
   * Typical aura without headache;
   * Familial Hemiplegic Migraine (FHM);
   * Sporadic Hemiplegic Migraine;
   * Basilar type Migraine;
4. Any laboratorial finding that the Investigator consider a risk to the subject of the study;
5. Hypersensitivity to the drug components, during the study;
6. Women in pregnancy or nursing period;
7. Women in reproductive age who do not agree to use contraception acceptable [oral contraceptives, injectable contraceptives, intrauterine device (IUD), hormonal implants, barrier methods, hormonal patch and tubal ligation]; other than surgically sterile (bilateral oophorectomy or hysterectomy), postmenopausal for at least one (01) years or sexual abstinence;
8. Inability to understand and answer to the functional categorical scale of the study, diary of symptoms, and not having accompanying to assist him/her;
9. History of abuse, according to the principal investigator, of the alcohol, opioids, barbiturates, benzodiazepines and illicit drugs in the last 02 years, or abuse of drugs for headache including ergotamines or narcotics in the last 03 months;
10. Subjects with prolonged hypotension, shock, sepsis, pheochromocytoma, hemorrhage, mechanical obstruction or perforation of the gastrointestinal tract;
11. Subjects with history of epilepsy or presence of psychiatric illness of any kind, in the opinion of the investigator, that may interfere with adherence to treatment;
12. Subjects with a malignant disease less than five years, or for more than five years, but without documentation about the remission/cure. As example: melanoma, leukemia, lymphoma, myeloproliferative diseases and renal cell carcinoma of any length should be excluded. Exceptions: Subjects with basal cell skin cancers, squamous cell, and cervical cancer in situ may be eligible.
13. Subjects which uses a preventive treatment and changed the dose in the last 3 months before the screening visit (V0);
14. Subjects who have made an interruption in the prophylactic treatment, in the last 30 days prior to screening visit (V0);
15. Subjects with hepatic or renal failure;
16. Subjects in the research that has participated in clinical trial protocols in the last twelve (12) months (National Board of Health- Resolution 251 of 07 August 1997, Part III, sub-item J), unless the investigator considers that there may be a direct benefit to it;
17. Subjects who are in prohibited medication as described in item 10.2 of the Protocol.
18. Subjects with previous diagnosis of uncontrolled hypertension;
19. Subjects with history of peripheral vascular disease; acute myocardial infarction, angina pectoris and other ischemic heart disease;
20. Subjects who have allergy to pyrazolones (eg phenazone, propyphenazone) or pyrazolidines (eg phenylbutazone,oxyphenbutazone) or who have submitted agranulocytosis in relation to any of these medicines;
21. Subjects with history of metabolic disorders such as porphyria and congenital deficiency of glucose-6-phosphate dehydrogenase;
22. Subjects with history of alteration in the bone marrow function or hematopoietic system diseases;
23. Subjects with history of bronchospasm or other allergic reactions (rhinitis, urticaria, angioedema) induced by aspirin, acetaminophen, or other anti-inflammatory medications.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy and non-inferiority of Cefaliv® compared to Neosaldina® in pain relief | 2 Hours
  The evaluation will be measured by the absolute variation of VAS (0 mm no pain - 100 mm pain as bad as can be) 2 hours after taking the medication, without taking any rescue medication.

SECONDARY OUTCOMES:
The remission of the pain after use of the investigational product, without use of a rescue medication; | 2 and 4 hours after taking the medication
  Proportion of participants with pain remission in 2 hours and 4 hours after the use of the investigational product, in the first migraine attack with mild or moderate pain, with remission defined as no pain (0) in categorical scale debilitating functional and behavioral (4 point-scale), without use of a rescue medication;
The relief of pain after use of the investigational product, without use of a rescue medication; | 2 and 4 hours after taking the medication
  Proportion of participants with pain relief in 2 hours and 4 hours after the use of the investigational product, in the first migraine attack with mild or moderate pain,and is considered the relief reduction of at least 01 point in pain intensity from baseline, according to functional and behavioral debilitating categorical scale without use of a rescue medication;
Proportion of participants with pain relief maintenance during the period 4-24 hours after use of the investigational product, the first migraine attack with mild or moderate pain | 4 to 24 hours after taking the medication
  The maintenance will be observed if the relief reached the first 4 hours will remain at 24 hours after use of the investigational product, according to functional and behavioral debilitating categorical scale (4 point scale) without use of a rescue medication during this period;
Need for use of a rescue medication. | 2 to 24 hours after taking the experimental drug
  Proportion of participants who use at least once a rescue medication in the period 2-24 hours after use of the investigational product.
The proportion of subjects with no symptoms of Nausea / vomiting and photophobia / phonophobia | 2 to 4 hours after taking the medication
  Free of photophobia, phonophobia, nausea and vomiting response rate symptoms 2 and 4 hours after use of the investigational product, the first with migraine pain of mild to moderate intensity, defined as the proportion of subjects with no symptoms of both among the participants have at least one symptom at baseline of migraine without use of a rescue medication during this period.

CONTACTS AND LOCATIONS:
Locations (1):
- Ache Laboratorios Farmaceuticos, Guarulhos, São Paulo, Brazil